CLINICAL TRIAL: NCT07313878
Title: Evaluation of Acute and Chronic Nephrotoxicity in Acute Lymphatic Leukemia Patients Using Ultrasound Localization Microscopy
Acronym: HEALED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HEALED-ULM
Record Dates: First submitted 2025-11-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukaemias (ALL); Long Term Follow-Up
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early therapeutic effects (Experimental): * Diagnosed acute lymphatic leukemia
  * Treatment day < 50 according to therapy protocol / no administration of CPM before first examination
  * From 3 years to < 18 years
  Interventions: Diagnostic Test: Ultrasound Localization Microscopy (ULM); Diagnostic Test: Blood sample; Diagnostic Test: Urinanalysis; Diagnostic Test: Renal sonography
- Late therapeutic effects (Experimental): * Diagnosed acute lymphatic leukemia
  * Completed oncological treatment
  * From 3 years to < 18 years
  Interventions: Diagnostic Test: Ultrasound Localization Microscopy (ULM); Diagnostic Test: Blood sample; Diagnostic Test: Urinanalysis; Diagnostic Test: Renal sonography

INTERVENTIONS:
Diagnostic Test: Ultrasound Localization Microscopy (ULM) — Single Examination: ULM of the kidney after application of a contrast medium (SonoVue®, intravenous).
  Arms: Early therapeutic effects
Diagnostic Test: Ultrasound Localization Microscopy (ULM) — ULM of the kidney after application of a contrast medium (SonoVue®, intravenous) at two different time points:
  Timepoint 1: Before initiation of therapy, latest day 50 before 1st high-dose methotrexate or cyclophosphamide.
  Timepoint 2: After termination of intensive treatment (after 6-9 months).
  Arms: Late therapeutic effects
Diagnostic Test: Blood sample — Blood draw (including BB, Diff, Glucose, Na, K, Cl, Ca, LDH, Crea, Cystatin C, Uric Acid, CRP, Albumin, Ferritin, Total Protein) through venous access.
  Arms: Early therapeutic effects
Diagnostic Test: Blood sample — Blood draw (including BB, Diff, Glucose, Na, K, Cl, Ca, LDH, Crea, Cystatin C, Uric Acid, CRP, Albumin, Ferritin, Total Protein) through venous access at Timepoint 1 and 2.
  Arms: Late therapeutic effects
Diagnostic Test: Urinanalysis — Examination of urine for erythrocytes, leukocytes, pH value, nitrite, protein, blood, and electrolytes.
  Arms: Early therapeutic effects
Diagnostic Test: Urinanalysis — Examination of urine for erythrocytes, leukocytes, pH value, nitrite, protein, blood, and electrolytes at Timepoint 1 and Timepoint 2.
  Arms: Late therapeutic effects
Diagnostic Test: Renal sonography — Renal sonography including resistance index (RI), Doppler signal, flow velocity, and others.
  Arms: Early therapeutic effects
Diagnostic Test: Renal sonography — Renal sonography including resistance index (RI), Doppler signal, flow velocity, and others at time point 1 and time point 2.
  Arms: Late therapeutic effects

SUMMARY:
With increasing survival rates in pediatric oncology, reports of long-term side effects persisting decades after treatment are also rising. Clinically evident nephropathies occur in about 5.5% of survivors more than five years after therapy. Chemotherapeutic agents such as ifosfamide, cisplatin, and carboplatin, as well as kidney-directed treatments like radiation, surgery, or stem cell transplantation, increase this risk. Acute kidney injury has also been described in association with cyclophosphamide and high-dose methotrexate, which are used in the treatment of acute lymphoblastic leukemia (ALL). Studies show a high prevalence of albuminuria (around 14.5% of childhood cancer survivors), an early marker of kidney damage, while standard parameters like creatinine often become abnormal only at later stages.

Leukemia survivors suffer from vascular late effects caused by persistent endothelial damage triggered by cancer therapies such as anthracyclines, cyclophosphamide, and asparaginase, which increase inflammation and thrombosis risk. These vascular changes may also contribute to kidney injury.

ULM is a high-resolution ultrasound technique that uses microbubbles to visualize the microvasculature and resolve dynamic blood flow changes with a resolution beyond the diffraction limit. ULM is independent of kidney or liver function, has been applied in various organs, and was recently used for the first time to visualize glomeruli-the smallest functional units of the kidney-in humans. This method enables early detection of glomerular injury as a consequence of vascular damage, even before albuminuria appears, potentially allowing earlier adaptation of follow-up and initiation of treatment.

This pilot project focuses on survivors of ALL, as they are the largest and best studied pediatric cancer patient group also regarding late effects and, therefore, a sufficient number of individuals can be expected for his monocentric approach. Vascular functional impairment of the kidney could be detected at an early stage and the follow-up structures and measures such as the early use of nephroprotective drugs could be adapted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed acute lymphatic leukemia
* From 3 years to < 18 years
* completed oncological treatment or treatment day < 50 according to therapy protocol and no administration of CPM before first examination.

Exclusion Criteria:

* Known allergic disposition to SonoVue / other contrast agents
* Tattoo in the area of the examination field
* Pregnancy
* Breastfeeding mothers
* Contraindication for the use of Sonovue
* Critical condition
* Known clinically evident renal impairment

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
CEUS Measurement 1 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Peak enhancement (PE)
CEUS Measurement 2 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Wash-in area under the curve (WIAUC)
CEUS Measurement 3 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Wash-in perfusion index (WiPI)
CEUS Measurement 4 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Wash-in rate (WIR)
CEUS Measurement 5 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Wash-out under the curve (WoAUC)
CEUS Measurement 6 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Wash-in and wash-out under the curve (WiWoAUC)
CEUS Measurement 7 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Wash-out rate (WoR)
CEUS Measurement 8 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Time to peak (TTP)
CEUS Measurement 9 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Rise time (RT)
CEUS Measurement 10 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Mean transit time (local) (mTTI)
CEUS Measurement 11 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Fall time (FT)
CEUS Measurement 12 | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Peak enhancement (PE)

SECONDARY OUTCOMES:
Blood Count | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Complete blood count with number of red and white blood cells and platelets per µl
Urine status | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Measurement of proteinuria in mg/l with protein differentiation
RI | Measurement of proteinuria with protein differentiation
  Resistance index (Sonography)
Flow velocity | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Flow velocity in Doppler Signal (Sonography)
Weigth | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Weigth of the participant in kilograms
Height | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Height of the participant in meters
BP | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Measurement of systolic, diastolic and mean blood pressure in mmHg
Electrolytes | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Concentration of serum electrolytes (Na, K, Cl, Mg, P) in mmol/L.
Creatinin and urea level | Study arm early therapeutic effects: Baseline before day 50 of the therapy and follow up after completion of intensive chemotherapy Study arm late therapeutic effects: Baseline at a single-time point in oncological follow-up care
  Serum Creatinin and urea level in mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics and Adolescent Medicine, Erlangen, Baveria, Germany

IPD SHARING:
Plan to Share IPD: Yes
The raw, individual and identifiable patient data are protected and are not available due to data privacy laws. Further data sets are planned to be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request as follows:
  Individual participant data will not be available Study Protocol and Statistical Analysis Plan will be available The data will be available beginning 9 months and ending 36 months following article publication.
  The data will be available to researchers who provide a methodologically sound proposal.
  The data will be available for individual participant data meta-analysis, only. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at https://www.uk-erlangen.de.
  Restrictions may apply due to patient privacy and the General Data Protection Regulation.

DOCUMENTS (1):
  • Study Protocol (2025-09-02): https://cdn.clinicaltrials.gov/large-docs/78/NCT07313878/Prot_000.pdf